CLINICAL TRIAL: NCT03056586
Title: The Recurrence Rate of Genital Prolapse Post Repair With the Use of PESSARY for One Month Post Operative
Brief Title: The Effect of Pessary Post Vaginal Prolapse Repair, for One Month, to Reduce the Recurrence Rate of Prolapse
Acronym: pfgp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Klein zvi, Head of urogynecology unit, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0188-16-MMC
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Use of Pessary Reduce the Number of Prolapse Recurrence; Uterine Prolapse; Cystocele; Rectocele
MeSH Terms: conditions — Uterine Prolapse; Cystocele; Rectocele | interventions — Pessaries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1. study group (Experimental): 100 patients who agree to participate in the study, will be operate according to our protocol for pelvic organ prolapse. At the end of the operation a vaginal pessary will be inserted and suture to the vaginal walls for a 4 week period.
  Follow-up will be after 3, 6, and 12 month period.
  Interventions: Device: vaginal pessary
- 2. control (No Intervention): 100 Women who will refuse to participate in the study, will agree to be follow-up by our team for 3, 6, and 12 month post operative.

INTERVENTIONS:
Device: vaginal pessary — A vaginal pessary will be inserted at the end of the operation, for genital prolapse, and will be sutured to the vaginal wall. The pessary will stay in the vagina for 4 weeks.
  Arms: 1. study group

SUMMARY:
Genital prolapse is a common complain. 30-40% of women will complain of uterine prolapse or cystocele or rectocele, or mixed. About half of them will require surgical repair for the prolapse, with or without hysterectomy. Of these patients about 30-40% will have recurrence of the prolapse, which in some cases requires second operation.

In this study the investigators want to investigate whether a vaginal pessary inserting in the end of the primary surgery, for 4 weeks, will reduce the recurrence rate.

DETAILED DESCRIPTION:
All patients going for vaginal surgery for genital prolapse, stage 3-4, with cystocele, rectocele or uterine cervix prominent from the vagina. These patients, after signing an informed consent, a vaginal pessary will insert at the end of the operation and will stay for 4 weeks post-op.

After 4 weeks the pessary will be removed, and the patient will followed for 2 years, for recurrence of prolapse.

ELIGIBILITY:
Inclusion Criteria:

* all healthy patients with genital prolapse grade 3-4, going for vaginal surgery
* age 30-80years

Exclusion Criteria:

* patients with pelvic inflammatory disease
* patients after pelvic irradiation
* large vaginal erosion
* vaginal bleeding uncontrolled or undiagnosed
* patients going for surgery with mesh

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 100 (Estimated)
Dates: Start 2017-03-20 (Estimated); Primary Completion 2018-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Reduction of recurrence rate of vaginal prolapse, post vaginal surgery repair. | 24 month
  The investigators hope to see a low percentage of prolapse recurrence in the study (pessary) group, comparing to the control (no pessary) group